CLINICAL TRIAL: NCT00435071
Title: The Effect of Surgical Incision Size on Carpal Tunnel Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator initiated suspension to focus on other studies.
Sponsor: Vanderbilt University (Other)
Responsible Party: Dr. Donald Lee, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 061043
Record Dates: First submitted 2007-02-12; First posted 2007-02-14 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-02

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Procedure: Carpal Tunnel Release Surgery
- 2 (Active Comparator)
  Interventions: Procedure: Carpal tunnel release surgery

INTERVENTIONS:
Procedure: Carpal Tunnel Release Surgery — Patient will have large incision size during carpal tunnel release surgery.
  Arms: 1
Procedure: Carpal tunnel release surgery — Patient will have a small incision size during carpal tunnel release surgery.
  Arms: 2

SUMMARY:
This study will investigate the postoperative recovery advantages from having a smaller incision to a larger incision.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing open carpal tunnel release will be included in this study.
* Patients must have clinical evidence of Carpal Tunnel Syndrome
* Patients must have positive EMG results

Patient selection factors include:

1. Ability and willingness to follow instructions
2. Patients who are able and willing to return for follow-up evaluations.
3. Patients of all races and genders.
4. Patients who are able to follow care instructions.

Exclusion Criteria:

* Patients less than 18 years old
* Patients unwillingly or unable to comply with a rehabilitation program for carpal tunnel release who indicate difficulty or inability to return for follow-up visits prescribed by the study protocol.
* Patients who qualify for inclusion in the study, but refuse consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Function questionnaires, pain assessment questionnaires, and clinical measurements will be used to determine the outcome of this study. | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Julie Daniels, Study Director — VUMC
Locations (1):
- Vanderbilt Orthopaedic Institute, Nashville, Tennessee, United States